CLINICAL TRIAL: NCT07176637
Title: A-B-C Program: a Brief Intervention to Promote an Active Lifestyle by Addressing Behavioral Economics Cognitive Biases Among Sedentary Older Adults With Depressive Symptoms-a Randomized Controlled Trial
Brief Title: A-B-C Program for Sedentary Older Adults With Depressive Symptoms
Acronym: A-B-C
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 273; ROH-24-004 (Other Grant/Funding Number: Academic Health Sciences Centre (AHSC) Alternative Funding Plan (AFP) Innovation Fund)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Sedentary Older Adults; Sedentariness and Well-being; Sedentary; Aging
Keywords: sedentary older adults; depressive symptoms; behavioural economics; A-B-C Program; physical activity; decision making; automatic thoughts; cognitive biases
MeSH Terms: conditions — Sedentary Behavior; Depression; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-B-C Group (Experimental): The intervention group will be led by Dr. Klil-Drori, a staff academic psychiatrist in the Geriatric Department at The Royal Ottawa Mental Health Centre. Dr. Klil-Drori completed clinical and research postdoctoral fellowships at McGill University and the University of Toronto, and developed the "A-B-C" program. The "A-B-C" program is a structured group intervention that meets twice weekly for four weeks, with each session lasting 60 minutes. Small groups of five participants will be facilitated by Dr. Klil-Drori. The program covers topics such as automatic thoughts and their associated emotions, common cognitive distortions (or cognitive biases), and how these influence decision-making and behaviour. Concepts introduced during sessions will be reinforced through structured group discussions and daily home practice assignments. The full outline for the A-B-C program, and the program journal can be found in 'Other Documents'.
  Interventions: Behavioral: A-B-C Program
- Physical activity education (Active Comparator): The control group will serve as an sham active comparator, designed to control for group format, scheduled sessions, and social interaction. The agenda for the control group was designed to specifically function as a control to compare the A-B-C program. These participants will also attend twice-weekly 60-minute sessions over four weeks, focusing on educational content about the health benefits of physical activity and current physical activity guidelines.
  The difference between the two interventions is that the control program is strictly educational, whereas the A-B-C program focuses on challenging cognitive biases that change decision making related to physical activity. To reiterate, the control program simply provides education on the effects of physical activity with physiological evidence.
  Interventions: Other: Physical Activity Educational Program

INTERVENTIONS:
Behavioral: A-B-C Program — The purpose of this study is to assess the effectiveness of the 4-week "A-B-C" program in implementing and maintaining daily PA. We will explore outcomes for the effectiveness of the program, on (1) increasing the weekly duration of PA, and (2) reducing baseline depressive symptoms and other mental health outcomes among sedentary older adults with depressive symptoms at baseline. Specifically, we will evaluate the change in depressive symptoms, stress, and self-esteem from baseline, at the end of the 4-week intervention, and after additional 4 weeks from the end of the intervention (at follow-up). The intervention will be 4 weeks overall, with total of 8 sessions: the duration of each session will be 60 minutes each, and the frequency will be twice weekly for 4 weeks.
  Arms: A-B-C Group
Other: Physical Activity Educational Program — The control group will serve as an sham active comparator, designed to control for group format, scheduled sessions, and social interaction. The agenda for the control group was designed to specifically function as a control to compare the A-B-C program. These participants will also attend twice-weekly 60-minute sessions over four weeks, focusing on educational content about the health benefits of physical activity and current physical activity guidelines.
  The difference between the two interventions is that the control program is strictly educational, whereas the A-B-C program focuses on challenging cognitive biases that change decision making related to physical activity. To reiterate, the control program simply provides education on the effects of physical activity with physiological evidence.
  Arms: Physical activity education

SUMMARY:
The importance and benefits of leading a physically active lifestyle have been long studied. Examples of the multiple advantages from physical activity are improved health of the heart and brain, having a more independent living and better quality of life. However, it is known that for many people, being active is challenging: physical activity is commonly viewed as a burden or inconvenience. In this study we will explore how some common everyday thoughts are hurdles to becoming physically active. We will discover ways to overcome this by using concepts from a field called "behavioral economics" that explains how we make decisions. The purpose of the program is to support participants in being more physically active. The study program is a newly developed way to overcome the intuitive preference for being sedentary. The experimental groups will learn simple ways to overcome expected hurdles in making decisions related to physical activity (the newly developed program), and the control groups will learn about the health benefits of physical activity and the health guidelines (the common practice today). We will compare the effectiveness of the newly developed intervention in promoting an active lifestyle, compared to the common practice today, of providing the knowledge and the recommended guidelines. The program in the study will be in small groups of 5-10 participants that will meet at The Royal for 60 minutes, twice a week, for 4 weeks.

DETAILED DESCRIPTION:
The lifetime prevalence of depression in Canada is approximately 11% in the general population (Patten et al., 2016). Additionally, depression is a leading cause for disability and carries a high cost to the Canadian economy, estimated over $50 billion CAD annually (Mental Health Commission of Canada, 2013). Cost-effective preventive measures for depression are required. Among the preventive methods, there is growing evidence on the advantages of physical activity (PA) for improving brain health, reducing depressive symptoms and preventing cognitive decline (Iso-Markku et al., 2024; Schuch et al., 2016). Suggested mechanisms in which PA contributes to brain health are enhanced neural metabolism, increased cerebrovascular flow, and improved neuroplasticity, in addition to better release of neurotrophic factors and neurotransmitters which contribute to improving depressive symptoms, maintaining cognitive reserve and preventing neurovascular and neurodegenerative conditions (Guan et al., 2024; Umegaki et al., 2021).

Conversely, physical inactivity is a significant risk factor for morbidity and mortality, including risk for depression (Kamphuis et al., 2007). In addition, physical inactivity carries a high economic burden: the total healthcare costs of physical inactivity in Canada is $9.3 billion CAD annually (Janssen, 2012). Moreover, the prevalence of physical inactivity significantly increases with age. In addition to the high prevalence of inactivity in the general population, depression is an independent disabling condition that frequently presents with reduced energy, low motivation, and decreased levels of physical activity. Therefore, people with depression are even more commonly inactive. However, there is a positive association between PA and reduced depression: a recent systematic review and meta-analysis by Pearce and colleagues (2022), explored the association between PA and the risk of depression among adults. This meta-analysis included 15 prospective cohort studies and 191,130 participants in prospective studies with a minimum of 3-years follow-up; it showed a significant improvement in depressive symptoms in adults who engaged in PA even in low doses, below the recommended dose in the PA health guidelines, compared to adults who reported no PA (Pearce et al., 2022). The suggested impact of PA at any dose on reduced depressive symptoms may suggest the importance of encouraging patients to be physically active even at lower doses than the PA health guidelines.

The Active Lifestyle using Behavioral Economics based Cognitive Biases (A-B-C) study program was recently developed with purpose to efficiently implement and maintain an active lifestyle. It is unique due to the aim of identifying barriers in maintaining a physically active lifestyle, and targeting the process of decision making, with focus on Behavioral Economics (B/E) concepts, as opposed to behavior change or behavioral activation. It integrates concepts from B/E, Cognitive Behavioral Therapy (CBT) and Logotherapy, in a 4-week program aimed at promoting an active lifestyle among sedentary adults with depressive symptoms. In this pilot study, we expect that this brief 4-week program will be effective in (1) promoting PA and (2) reducing depressive symptoms.

Participation in the A-B-C program carries minimal risk. Potential risks include psychological discomfort when discussing cognitive patterns or depressive symptoms, and mild physical discomfort from increased activity. However, these risks are expected to be low and will be mitigated by careful facilitation, screening, and referral mechanisms. Expected benefits include reduced depressive symptoms, increased motivation for physical activity, and improved cognitive-emotional awareness.

The A-B-C program is delivered in-person by a trained psychiatrist and includes twice-weekly, 60-minute sessions over four weeks. Measures include validated self-report questionnaires assessing depressive symptoms (e.g., PHQ-9), stress (PSS-10) and self-esteem (RSE), and self-reported logs of physical activity. Participants in the intervention also complete daily home assignments to reinforce session content. Follow-up assessments are conducted at baseline, post-intervention, and 3, 6, 9, and 12 months. The control group receives an active comparator intervention consisting of general educational sessions about physical activity benefits and guidelines, matched for frequency, duration, and format. While the A-B-C program is a novel intervention, it draws upon evidence-based components validated in other contexts: behavioral economics interventions in health behavior change (Loewenstein et al., 2007), CBT for depression (Beck, 1979), and motivational programs using logotherapy principles (Frankl, 1985). No previous trials have tested this specific synthesis; this pilot study aims to establish preliminary efficacy.

The purpose of this study is to assess the effectiveness of the 4-week "A-B-C" program in implementing and maintaining daily PA. We will explore outcomes for the effectiveness of the program, on (1) increasing the weekly duration of PA, and (2) reducing baseline depressive symptoms and other mental health outcomes among sedentary older adults with depressive symptoms at baseline. Specifically, we will evaluate the change in depressive symptoms, stress, and self-esteem from baseline, at the end of the 4-week intervention, and after additional 4 weeks from the end of the intervention (at follow-up). The intervention will be 4 weeks overall, with total of 8 sessions: the duration of each session will be 60 minutes each, and the frequency will be twice weekly for 4 weeks. The purpose of the study intervention is to explore the process of decision-making and automatic thoughts that are related to planning PA, and modify cognitive biases that may prevent a person from engaging in PA. Following participation in the study, we will conduct qualitative semi-structured interviews to establish a better understanding of the participants' subjective experience in the study, which will provide additional insight and may also suggest modifications to the program.

We hypothesize that the A-B-C Program will increase physical activity, reduce depressive symptoms, improve self-esteem, and reduce stress.

The objectives of the study are to determine the relative effectiveness of the program on the following measures, at 4 weeks from baseline (post-intervention) and 3, 6, 9, and 12 months post-intervention (follow-up points) compared to baseline and to the control group:

1. Weekly dose of physical activity: daily duration and intensity of physical activity, measured by self-report in the daily program journal.
2. Depressive symptoms, as measured by the PHQ-9
3. Self-esteem, measured by the Rosenberg Self-Esteem (RSE) scale
4. Stress, measured by the Perceived-Stress-Scale (PSS)

ELIGIBILITY:
Inclusion Criteria:

* 1. All sex and gender inclusive 2. Age 65 and over 3. Cognitive telephone screening via the 20-point Tele-MoCA with a score of 16 or higher.

  4. Score on the PHQ-9 is between 2-14. 5. The participant agrees to attend all the meetings for the duration of the study, and to practice home assignments.

  6. Adequate command of English to be able to participate in the group sessions. 7. Current weekly duration of exercise* ≤60 minutes/week. (*Exercise: a specific type of physical activity [PA], which is structured, and has the intention of improving either health or fitness. Exercise differs from PA, which includes any physical effort, however without the intention of improving health or fitness [e.g., driving, cleaning, standing, etc. are examples for PA, not exercise]) 8. Participants have interest in increasing their weekly time of physical activity, and willingness to practice skills learned during the program.

  9. Agree to participate in any of the study groups according to a randomized allocation.

Exclusion Criteria:

* 1. Acute medical condition that requires treatment. 2. Existing medical conditions that contra-indicate or limit physical activity (e.g., post-surgery, recurrent falls, etc.) 3. Unstable psychiatric condition that requires acute care. 4. Current use of psychoactive medication that might compromise balance or induce risk when performing physical activity (e.g., high dose of sedative medications) 5. Current use of recreational drug use (must be free of substance use for 12 months).

  6. Patients currently involved in routine intensive exercise* > 1 hour/ week. 7. Lack of interest to increase their daily time of physical activity 8. Refuse to participate in any of the study groups according to a randomized allocation.

  9. PHQ-9 score less than 2, or greater than 14.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Daily dose of PA | From enrollment to the end of treatment at 4 weeks (post-intervention); every 3 months up to 12 months post-intervention.
  Daily dose of PA (intensity, duration) - will be self-reported and recorded participants in their daily program journals.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | From enrollment to the end of treatment at 4 weeks (post-intervention); every 3 months up to 12 months post-intervention.
  This is a validated 9-item questionnaire that is used to measure depressive symptoms. A clinically significant improvement in depressive symptoms will be defined by a finding of a statistically significant change of the PHQ-9 score at the time of assessment, compared to the PHQ-9 score at baseline, of each individual. The study population is defined with depressive symptoms: one of the inclusion criteria for the study is a minimum PHQ-9 score of 2 at baseline and a maximum score is 14.
Rosenberg Self-Esteem Scale (RSE) | From enrollment to the end of treatment at 4 weeks (post-intervention); every 3 months up to 12 months post-intervention.
  The scale is a ten-item Likert scale with items answered on a four-point scale - from strongly agree to strongly disagree. The higher the score, the higher the self-esteem. A successful measurement is defined as a minimum increase of 10% on the score of RSE at baseline.
Perceived Stress Scale | From enrollment to the end of treatment at 4 weeks (post-intervention); every 3 months up to 12 months post-intervention.
  4. The Perceived Stress Scale (PSS-10) is a 10-item scale that will be used to measure stress, inquiring how participants felt in the past month and the degree to which life events were experienced and appraised as stressful, with responses ranging from 0 (never) to 4 (very often).

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.